CLINICAL TRIAL: NCT06301087
Title: An Observational Cross-Sectional Study of Early Detection of 5 Neurodevelopmental Disorders of Children and Prevention of Postnatal Depression by Mobile Health App
Brief Title: Early Detection Neurodevelopmental Disorders of Children and Prevention of Postnatal Depression by Mobile Health App
Status: Completed | Type: Observational
Sponsor: Weprom (Other)
Collaborators: Kelindi (Industry)
Responsible Party: Sponsor
Other Study IDs: WP-2024-01
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Development, Child; Postnatal Depression
Keywords: early detection; neurodevelopmental disorders; postnatal depression; mHealth; real-world study; smartphone
MeSH Terms: conditions — Depression, Postpartum; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- users: users of the web-application
  Interventions: Device: Web Application

INTERVENTIONS:
Device: Web Application — web application for monitoring children's development and postnatal depression of mothers
  Other Names: MALO

SUMMARY:
The goal of this observational study is to confirm the impact of using this app adapted to be more specific for screening for 5 neurodevelopmental disorders and to evaluate the mothers' support program on the incidence of postpartum depression in of young parents with a minimum of 1 child under 10 years of age at the time of inclusion and using Malo on a regular basis. The main questions it aims to answer are :

* the median age of possible neurodevelopmental disorders notification of infants
* the median time of the mothers' postnatal depression notifications after childbirth subsequently to the support and prevention program Participants will agree with use of their data

ELIGIBILITY:
Inclusion Criteria:

* Youg parent with a minimum of 1 child under 10 years
* User of the app (downloaded)
* Having given informed consent (in-app)

Exclusion Criteria:

* none

Max Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population will include the first 50,000 users of the application who consent to the use of their data for this assessment
  young parent withe a minimum of 1 child under 10 years matching the criteria and agreeing to participate
Sampling Method: Non-Probability Sample
Enrollment: 55618 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Time to neurodevelopment desorder diagnostic | 20 months
  Number of days between birth and notification of possible neurodevelopment desorder notification

SECONDARY OUTCOMES:
User's satisfaction | 20 months
  Home made qualitatif satisfaction questionnaire
Relevance of the neurodevelopmental desorder notification | 20 months
  Parent's feedback for physician's opinion after notification
Rate of mothers'postnal depression | 20 months
  Number of mothers with grade 2 ou 3 at adapted Edimbourg postnatal depression scale
Time of mothers'postnatal depression | 7 months
  Number of days between Edimbourg postnatal depression scale grade 2 or 3 and childbirth (score 0 to 30 a higher score indicates a worse condition)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice DENIS, Principal Investigator — Kelindi
Locations (1):
- ILC, Le Mans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denis F, Le Goff F, Desbois M, Gepner A, Feliciano G, Silber D, Zeitoun JD, Assuied GP. Early Detection of 5 Neurodevelopmental Disorders of Children and Prevention of Postnatal Depression With a Mobile Health App: Observational Cross-Sectional Study. JMIR Public Health Surveill. 2024 Jun 18;10:e58565. doi: 10.2196/58565. PMID 38888952